CLINICAL TRIAL: NCT06902506
Title: Exploring the Effects of Sonic Augmentation Technology in Music on Feelings and Biobehavioral State
Brief Title: Exploring the Effects of Sonic Augmentation Technology in Music
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Keeping the study open for future recruitment.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB202500241
Record Dates: First submitted 2025-03-18; First posted 2025-03-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Sonic Augmentation Technology
Keywords: Polyvagal Theory; Relaxation; Autonomic Reactivity

STUDY DESIGN:
Intervention Model Description: Phase 1: Participants will be randomly assigned to the augmented or non-augmented music group. Both groups will complete an online pre-music survey. Following the 15-minutes of music, participants will complete an online post-music survey.
  Phase 2: Participants will complete an online pre-music survey. Then, they will listen to 15-minutes of augmented music. Following the 15-minutes of music, participants will complete an online post-music survey.
Who Masked: Participant
Masking Description: Phase 1 ONLY: Participants will be randomly assigned to either the augmented group or the non-augmented group. The participant will be blinded to the group they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Group (Experimental): Phase 1 & 2: Participants will first complete the pre-music survey. They will then listen to 15 minutes of augmented music. Afterward, participants will complete the post-music survey.
  Interventions: Behavioral: Augmented Music
- Non-augmented Group (Active Comparator): Phase 1 ONLY: Participants will first complete the pre-music survey. They will then listen to 15-minutes of the same musical theme without the augmentation. Afterward, participants will complete the post-music survey.
  Interventions: Behavioral: Non-augmented Music

INTERVENTIONS:
Behavioral: Augmented Music — Phase 1 & 2: The music is augmented by embedding the natural rhythms of bodily functions (e.g. breathing, heart rate variability, vascular tone, etc) that signal the body to calm.
  Arms: Augmented Group
Behavioral: Non-augmented Music — Phase 1 ONLY: Same melodic theme without the augmentation.
  Arms: Non-augmented Group

SUMMARY:
Brief Summary:

It is the specific intent of this proposal to experimentally explore the possible benefits and mechanisms through which Sonic Augmentation Technology in music can influence emotional health, embodiment, and autonomic functioning. The main goals of the study are:

* To examine the immediate effects of listening to the music.
* To identify individual characteristics that influence the effectiveness of listening to the music.
* Phase 1 ONLY: To examine whether the participants who received the augmented theme reported more improvements than the participants who received the non-augmented theme.

Participants will be asked to attend a scheduled online Zoom meeting where they will:

* Listen to 15-minutes of music
* Complete a pre-music and post-music online survey
* Phase 1 ONLY: Attend the lecture/discussion with Dr. Porges and Anthony Gorry on theory and science underlying sonic augmentation technology and the experiences it aims to evoke.

DETAILED DESCRIPTION:
Detailed Description:

It is the specific intent of this proposal to experimentally explore the possible benefits and mechanisms through which Sonic Augmentation Technology (SAT) in music can influence emotional health, embodiment, and autonomic functioning. This will be accomplished by our team by using well-validated self-report measures of mental health and autonomic reactivity.

Specific Aims:

Specific Aim 1: To examine the immediate effects of SAT in music

•The researchers will explore whether SAT in music leads to improvements in the functioning.

Specific Aim 2: To identify individual characteristics that influence the effectiveness of listening to the music.

* The researchers will explore the impact of specific vulnerability and resiliency factors (e.g., prior mental and medical adversity) on how well participants benefit from listening to the music.
* The researchers will explore the impact of wearing headphones on how well participants benefit from listening to the music.

Phase 1 Experimental design:

Participants will be randomly assigned to either a Sonic Augmentation Technology-enhanced music condition or a control condition featuring the same musical theme without the enhancement. Participants will be asked to attend one virtual session via Zoom where they will:

* Listen to 15-minutes of music
* Complete a pre-music and post-music online survey
* Attend the lecture/discussion with Dr. Porges and Anthony Gorry on theory and science underlying sonic augmentation technology and the experiences it aims to evoke.

Phase 2 Experimental design:

Participants will be asked to attend one virtual session via Zoom where they will:

* Listen to 15-minutes of music
* Complete a pre-music and post-music online survey
* At a later date, participants will be offered the opportunity to attend an optional meeting where results will be disseminated, and Dr. Stephen Porges will be offering insights into the theory and science underlying sonic augmentation technology and the experiences it aims to evoke.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 89
* Proficient in English

Exclusion Criteria:

* Under the age of 18
* Over the age of 89
* Limited English Proficiency

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Assessing the Impact of Autonomic Reactivity using the Body Perceptions Inventory Short Form | Baseline
  This 20-item measure is scored on a 5-point Likert scale (never = 1, occasionally = 2, sometimes = 3, usually = 4, always = 5). Items are summed to determine total autonomic reactivity score, with the higher scores indicating greater autonomic reactivity
Assessing the Impact of Adversity History | Baseline
  This measure assesses the impact of six types of traumatic experiences (childhood adverse experiences, childhood maltreatment, intimate partner maltreatment, other person maltreatment, life-threatening situations, sudden losses, and person health situations). Each item is scored on a 5-point Likert scale (did not occur = 0, occurred and no impact on my life = 1 to big impact on my life = 4). Items are summed to determine total impact scores.
Measuring Change in subjective feelings of calmness and autonomic state using the Benefits List | From baseline through study completion, an average of 65 minutes
  This 20-item measure, which assesses subjective feelings of calmness and autonomic state was created for this study. Each item is scored on a 7-point Likert scale (0 = Not at all, 3 = Somewhat, 6 = Extremely). Higher scores on the scale generally represent increased feelings of calmness and a more balanced autonomic state.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes P Dale, BS, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be available.